CLINICAL TRIAL: NCT04177875
Title: A Phase II, Prospective, Open-label Clinical Trial of Pre-Operative PD-1 Antibody (Toripalimab) + Chemoradiotherapy in Patients With Locally Advanced Esophageal Cancer
Brief Title: Neoadjuvant Chemoradiotherapy Combined With PD-1 Antibody in Locally Advanced Esophageal Cancer
Acronym: T+TP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2019]（S910）
Record Dates: First submitted 2019-10-30; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-05

CONDITIONS: Esophagus Cancer
Keywords: neoadjuvant therapy；pd-1 antibody combined with Chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Docetaxel; Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiation and pd-1 (Experimental): Subjects in Arm A receive 2 cycles of Docetaxel /Albumin-bound Paclitaxel + Cisplatin, for neoadjuvant therapy Neoadjuvant radiotherapy for 40Gy/20F
  Interventions: Drug: Teripalimab

INTERVENTIONS:
Drug: Teripalimab — Teripalimab Injection 240mg/6ml fixed dose (3mg/kg for patients weighing less than 40kg) ,injection on day 1, each infusion for 30min (no less than 60 minutes for the first injection); every 3 weeks. docetaxel dose was 75mg/m2, injection on day 1;Albumin-bound Paclitaxel (no anti-allergic treatment required), 260mg/m2, injection on day 1; Cisplatin was 75mg/m2, injected on day 1.A total of two treatment cycles.
  Other Names: Docetaxel /Albumin-bound Paclitaxel; Cisplatin

SUMMARY:
This study will evaluate the safety and feasibility of preoperative immune checkpoint therapy with concurrent Chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma. And this study will provide valuable information for further clinical trials of preoperative Teripalimab and other immune checkpoint therapy in esophageal cancer treatment.

DETAILED DESCRIPTION:
Esophageal cancer ranks the eighth most common cancer in Worldwide. And the third among men and the fifth among women in China, among which esophageal squamous cell carcinoma accounts for about 90%.

Neoadjuvant therapy for esophageal cancer is increasingly supported by evidence. However, the results of neoadjuvant therapy are not completely consistent. Most studies of neoadjuvant treatment data for esophageal cancer were obtained from western populations, where esophageal adenocarcinoma and esophagogastric junction adenocarcinoma were more common and the sample size was relatively small. According to the meta-analysis of the reported results of randomized controlled trials, concurrent chemoradiotherapy has a higher pathological complete response rate than chemotherapy alone as neoadjuvant therapy. However, the 3-year survival rate of neoadjuvant chemoradiotherapy only showed an advantage in patients with squamous cell carcinoma (56.8%vs42.8%), but no significant difference in patients with adenocarcinoma (46.3%vs41.0%). Pathological complete remission rate of esophageal cancer after neoadjuvant chemotherapy is relatively low.

It can be seen that positive expression of programmed death ligand-1 is more common in Esophageal squamous cell carcinoma, and programmed death ligand-1 tends to be overexpressed compared with adjacent normal epithelial cells. The later the T-stage of the tumor, the higher the positive expression rate. In addition, programmed death ligand-1 expression is significantly correlated with lymphatic metastasis. Therefore, programmed death ligand-1 expression can promote tumor progression. The recurrence rate of patients with programmed death ligand-1 expression is higher after treatment, and the postoperative complete pathological remission rate is lower in programmed death ligand-1 positive patients. In addition, positive programmed death ligand-1 expression also reduces the sensitivity of radiotherapy, which may be contributing factors to poor prognosis of patients with positive pd-l1 expression. It is worth mentioning that clinical treatment will affect the expression level of programmed death ligand-1 in esophageal cancer tissues. Neoadjuvant concurrent chemoradiotherapy can up-regulate the expression of programmed death ligand-1 in ESCC significantly, while neoadjuvant chemotherapy can down-regulate the expression of pd-L1. However, radiotherapy can up-regulate the expression level of programmed death ligand-1 in esophageal cancer cells, which is positively correlated with radiation dose, and the combination of anti-pd-L1 therapy and radiotherapy can lead to increased tumor cell lysis, which also indicates the importance of comprehensive treatment of tumor.

There are relatively few studies on the treatment of esophageal cancer with pd-1 / pd-L1 inhibitors. Keynote-059 enrolled 259 patients with advanced gastric or gastroesophageal junction cancer in the phase II clinical trial of Pembrolizumab, with an objective response rate of 11.6%, complete response rate of 2.3%, and median response duration of 8.4 months. Persistent objective response rates were observed in both programmed death ligand-1 positive and negative patients, and adverse reactions were tolerable.

The efficacy and safety of anti-pd-1 / pd-L1 therapy in the treatment of esophageal cancer still need a lot of clinical studies to further confirm. This study will evaluate the safety and feasibility of preoperative immune checkpoint therapy using pembrolizumab with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma. And this study will provide valuable information for further clinical trials of preoperative Teripalimab and other immune checkpoint therapy in esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70, male or female
* Locally advanced esophageal cancer diagnosed by pathology, Clinical tumor stage should be T2-3N0-1M0
* No previous chemoradiotherapy
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Demonstrate adequate organ function as defined below (excluding the use of any blood components and cytokines during the screening period)
* Absolute neutrophil count (ANC) ≥1.5*109 /L; Platelet ≥90*109/L; Hemoglobin ≥ 9 g/dL; Serum albumin≥3g/dL
* Bilirubin≤1.5 x ULN; ALT and AST≤2.5 ULN; Serum creatinine ≤1.5 x ULN or creatinine clearance ≥40mL/min
* Female subject must have taken reliable contraceptive measures of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. and be willing to use an appropriate method of contraception during the trial and 8 weeks after the last administration of the test drug. Male subject should agree to use appropriate contraceptive methods or to have been surgically sterilized during the trial and 8 weeks after the last administration of the test drug.
* Subjects voluntarily participated in this study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

* Any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitritis, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction);Subjects with vitiligo or who have had complete remission from childhood asthma without any intervention after adulthood may be included; Asthma requiring medical intervention with bronchodilators was not included. Those who have used other drugs in clinical trials to study drugs within 4 weeks before their first use;
* Severe allergic reaction to monoclonal antibody
* The number of neutrophils in peripheral blood was lower than 1500/mm3;
* There are clinical symptoms or diseases of the heart that are not well controlled, such as: A. heart failure above grade 2 by the Criteria of NYHA; B. unstable angina pectoris; C. myocardial infarction occurred within 1 year; D. Clinically meaningful supraventricular or ventricular arrhythmias require treatment or intervention;
* Has a previous radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy;
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). or Has known active Hepatitis B (e.g. HBV DNA≥ 2000IU/ml or copy number ≥104/ml;) or Hepatitis C (e.g. HCV antibody positive).
* According to the judgment of the researchers, the subjects have other factors that may cause the forced termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, severe laboratory examination abnormalities, accompanied by family or social factors, which may affect the safety of the subjects, or the collection of data and samples.
* The researchers determined patients with high risk of esophageal perforation or no potential surgical feasibility through endoscopic ultrasonography or imaging examination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response Rate (MPR) | 30 days after the second cycle of treatment(each cycle is 21 days)
  No more than 10% of tumor cells were found in neoadjuvant surgical specimens.
Objective Response Rate (ORR) | At the end of cycles 2(each cycle is 21 days)
  Based on RECIST evaluation criteria, the proportion of patients with complete ORR was defined as the percentage of patients having a complete response or a partial response to protocol treatment. Objective response will be measured by RECIST 1.1.

SECONDARY OUTCOMES:
2-year Disease-Free Survival Rate (24 months DFS) | 2 years
  The 2-year DFS rate was defined as the rate of progression or death due to disease recurrence within 2 years
Media Disease-free Survival (mDFS) | Up to 5 years
  The time at which disease progression or death due to disease progression occurred in 50% of patients
Media overall survival (mOS) | Up to 5 years
  The time of death occurred in 50% of patients
The incidence of adverse events and the incidence of severe adverse events（ grade 3-4) | 60 days after the end protocol treatment
  Safety will be evaluated for all treated patients using CTCAE V 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China